CLINICAL TRIAL: NCT04780620
Title: Addressing Parent-Adolescent Relationship Issues in the Treatment of Adolescent Depression: A Pilot Study
Brief Title: Group Intervention to Improve Parent-Adolescent Relationships
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Madison Aitken, Clinician Investigator at Cundill Centre for Child and Youth Depression; Psychologist in the Child, Youth and Emerging Adult Program, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 098-2020
Record Dates: First submitted 2021-03-01; First posted 2021-03-03 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Depression
Keywords: youth depression; adolescent depression; psychosocial intervention; parent-adolescent conflict
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research personnel involved in data collection will be blind to participants' treatment condition (single blind). In addition, coders for the interaction task and speech sample will be blind to treatment condition (intervention versus control) and measurement time point (baseline vs. posttreatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Intervention Group (Experimental): The parent intervention group will undergo 8 weekly, manualized group sessions, with between 6 and 10 parent participants. Sessions are structured and follow an agenda including check-in and review of home practice, discussion of a skill or strategy, and review and assignment of home practice. Group sessions are held weekly for 1.5 hours and include both didactic, discussion, and practice elements, as well as assigned home practice.
  Interventions: Other: Parent Intervention Group
- Usual Care Group (No Intervention): Parents in the usual care condition will be involved in their adolescent's care as is standard in our clinical program. With adolescent consent, parents are invited to participate in a single, 2-hour orientation session for parents/caregivers that provides information about depression, as well as the role of sleep, diet, and exercise in improving mood. Based on adolescent preference, parents can also attend regular psychiatric appointments with their adolescent, in which they will receive further information about depression and may receive and provide information about their adolescent's depression symptoms and response to psychosocial and pharmacological interventions. This control condition will allow us to determine whether the parent intervention is more effective than a relevant clinical alternative.

INTERVENTIONS:
Other: Parent Intervention Group — Parents will be involved in 8 weekly sessions.
  Arms: Parent Intervention Group

SUMMARY:
This pilot randomized control trial investigates whether a psychosocial intervention targeting parent-adolescent conflict is feasible and acceptable, in preparation for a future trial that will test whether the intervention can improve treatment outcomes for youth diagnosed with depression.

DETAILED DESCRIPTION:
Parent involvement in psychosocial interventions for youth diagnosed with internalizing disorders has been cited as a contributor to better outcomes for these youth, and parent components have been included in several evidence-based interventions for adolescent mental health problems. Additionally, youth experiencing mood and behaviour changes that come about as a result of a depressive episode can lead to frustrated/overprotective reactions from parents, which can contribute to worse outcomes for these adolescents. Interventions focused on addressing parent-adolescent conflict and reducing negative interactions can potentially support recovery from depression and reduce episode relapse. However, there is very little research on including parent components in psychosocial interventions specifically aimed at youth depression. This randomized control trial aims to fill this gap by randomizing parents of youth receiving treatment for depression into either 1) an 8-week virtual or in-person group parent intervention, or 2) usual care.

Participants will be parents or caregivers (for simplicity, the term "parent" is used to refer to parents or caregivers) of adolescents aged 13-18 with depression who are referred for outpatient services at a mental health research hospital in Toronto, Canada. Their adolescents will also participate in the study in order to provide multi-informant data; however, should adolescents decline to participate in the study, their parent will still be able to take part.

Parents will complete a combination of questionnaire and observationally coded measures at pre- and posttreatment, along with questionnaire measures at mid-treatment and 3 months follow-up. Adolescents will only complete questionnaire measures for all four time points.

ELIGIBILITY:
Inclusion Criteria:

* parent/caregiver of an adolescent aged 13-18 years
* the adolescent is referred for outpatient services at CAMH
* adolescent has significant depressive symptoms, having either: a) a self-reported score of 23 or higher on the Mood and Feelings Questionnaire; or b) a depression diagnosis based on the Kiddie-Schedule for Affective Disorders and Schizophrenia from the last 3 months
* parent or youth endorse problematic levels of conflict in their relationship, having either: a) a total score of 9 or greater on the adolescent version, or a total score of 11 or greater on the parent version, of the 20-item Conflict Behavior Questionnaire; or b) a rating of 2 or higher on item 2 or 3 (Item 2 "getting along with your mother/mother figure;" item 3 "getting along with your father/father figure") of the youth-report version of the Columbia Impairment Scale
* both parent and adolescent speak, read, and write English at a Grade 6 level or above

Exclusion Criteria:

* the adolescent's primary diagnosis is not depression, based on information in their health record
* the adolescent has been diagnosed with bipolar disorder (I or II), schizophrenia, moderate-severe eating disorder, moderate-severe substance use disorder, or an intellectual disability (as the clinical and family needs of these adolescents are not likely to be sufficiently addressed by a general group for parents of adolescents with depression), or requires immediate hospitalization for suicide risk
* the parent/caregiver does not consent to participate
* (specific only to the virtual format of the study) the parent is not comfortable communicating via email or using WebEx for virtual appointments (as the use of WebEx and email is required for study visits and for participation in the parent intervention)

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility Outcomes | 2 years (study duration)
  Feasibility defined as:
  * Participant recruitment rates, retention in the study, and completion of measures across time points
  * Parent satisfaction with the intervention
  * Parent attendance at the group and dropout from the group
  * Clinician fidelity to the intervention

SECONDARY OUTCOMES:
Parent Expressed Emotion | Pre-, mid- (4 weeks), and post-treatment (8 weeks), and at 3-month follow-up
  Parent report on the Family Questionnaire; Adolescent report on the Level of Expressed Emotion questionnaire; Observational coding of parent Five Minute Speech Sample
Parent Affective Responding | Pre-, mid- (4 weeks), and post-treatment (8 weeks), and at 3-month follow-up
  Parent and adolescent report on the Coping with Children's Negative Emotions Scale and the Responding to Adolescents' Happy Affect Scale
Parent-Adolescent Conflict | Pre-, mid- (4 weeks), and post-treatment (8 weeks), and at 3-month follow-up
  Parent and adolescent report on the Issues Checklist
Adolescent depression | Pre-, mid- (4 weeks), and post-treatment (8 weeks), and at 3-month follow-up
  Adolescent self-report on the Mood and Feelings Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Madison Aitken, Ph.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Sharing IPD has not currently been approved by our Research Ethics Board and would also require a data sharing agreement.